CLINICAL TRIAL: NCT04028089
Title: Nutritional Prevention of Gestational Diabetes Mellitus
Brief Title: Prevention of Gestational Diabetes
Acronym: NuPreGDM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 104/2019BO1
Record Dates: First submitted 2019-07-16; First posted 2019-07-22 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet Modification Group (Experimental)
  Interventions: Behavioral: Diet Modification Group
- Regular Diet Group (Other)
  Interventions: Other: Regular Diet Group

INTERVENTIONS:
Behavioral: Diet Modification Group — The diet modification group will receive diet counselling by an experienced dietician at least every four weeks throughout pregnancy starting in the first trimester. The dietary counselling will be guided by the individual glucose profiles obtained through flash glucose monitoring.
  Arms: Diet Modification Group
Other: Regular Diet Group — Participants of the "standard diet" will receive general diet counselling on one occasion at the onset of the study.
  Arms: Regular Diet Group

SUMMARY:
Pregnancy is a vulnerable period for both a mother and her developing child. The investigator hypothesizes that diet-induced glucose excursions in the pregnant mother are a key contributor to unfavourable brain development and epigenetic marks in the developing child. It is long known that metabolic conditions are influenced by maternal nutrition and that this can impact the unborn infant. The most prominent example is gestational diabetes (GDM). It is unclear at what point unfavourable changes in brain development occur during pregnancy. Unlike many previous trials, we plan to introduce healthy diet early in the first trimester. Comparative analyses of DNA methylation patterns in the offspring of women with or without GDM revealed preferentially methylated genes, particularly in pathways linked to metabolic diseases.

NuPreGDM is a randomized, controlled, open label intervention trail. The investigator aims to assess the effect of individual diet counselling combined with CGM compared to regular diet on glucose levels and postprandial glycemic excursions during an OGTT in pregnancy.

The investigator wants to assess the effect of dietary counselling combined with continuous glucose monitoring on GDM risk, glycaemia and pregnancy outcome, starting in the first trimester. The investigator further hypothesizes that improved glucose levels by a healthy diet will affect brain activity of the infant and prevent unfavourable epigenetic modifications.

The investigator plans to include 50 pregnant women within gestational week 4 and 14 after the last menstruation, with elevated risk for development of (GDM). Participants will be randomized 1:1 to either "diet modification group" (intervention) or to "standard diet group" (control). In the current trial, the investigator aims to modulate maternal metabolism with periodic personalized diet counselling on the basis of continuous glucose monitoring (CGM) compared to regular diet throughout pregnancy. The investigator propose that a reduction in glucose excursions in the mother will lead to a healthy environment for the developing child and prevent altered brain activity in utero, which will be assessed by fMEG (fetal magnetoencephalography) during a 75g OGTT in gestational week 28. The investigator further planned to examine child's leucocytes from cord blood to assess whether a healthy diet of the mother prevented epigenetic alterations due to improved maternal glycaemia, as exploratory endpoint. The development of blood sugar levels of the mother postpartum will be assessed by an further OGTT 6-12 weeks postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between gestational week 4 and 14 after the last menstruation (proof of b-human choriongonadotropin in urine or proof of pregnancy via ultrasound.)
* Pre-pregnancy overweight (pregravid BMI > = 27) or positive family history of type 2 diabetes or GDM in first-degree relatives or GDM in previous pregnancy or previous macrosomia (baby with birth weight > 4000 g) or advanced maternal age > = 40 years
* Ability to understand and voluntarily sign an informed consent document prior to any study related procedures.

Exclusion Criteria:

* Age < 18 years
* Multiple pregnancy
* Pre-pregnancy Diabetes mellitus
* Intake of medication that interferes with glucose-metabolism, such as glucose lowering or increasing drugs at inclusion visit (e.g. Steroids, Antidiabetics, Insulin, Metformin)
* Treatment with drugs with central nervous actions
* Chronic alcohol disease and drug abuse
* Pre-existing cardiac condition
* Mental disorder
* Weight loss >10% in the previous 6 months
* GFR < 60 ml/min/1.73 m2
* 2-fold increased transaminase levels in reference to the upper standard
* Any other (clinical) condition that would endanger participant's safety or question scientific success according to a physician's opinion.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-07-15 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Glycaemic excursion during an oral glucose tolerance test | gestational week (GW) 24 - 28
  The effect of a diet modification on glucose levels and postprandial glycemic excursions (AUC) during a 75g oral glucose tolerance test (OGTT) will be measured.

SECONDARY OUTCOMES:
Glucose variability | Gestational week 14,20, 28, 34 and one week postpartum
  The effect of diet modification during pregnancy on 24h glucose profiles and postprandial glycemic excursions (AUC) will be measured by flash glucose monitoring.
Maternal weight gain during pregnancy | Gestational week 14,20, 28, 34
  Body weight will be measured regularly during pregnancy.
Maternal insulin sensitivity | gestational week (GW) 24 - 28 and 6-12 weeks postpartum
  Whole body insulin sensitivity will be quantified from 5 point 75g oral glucose tolerance test.
Maternal insulin secretion | gestational week (GW) 24 - 28 and 6-12 weeks postpartum
  Insulin secretion will be quantified from 5 point 75g oral glucose tolerance test.
Fetal brain activity | Gestational week 28
  Fetal brain activity will be assessed by fMEG (fetal magnetoencephalography).
Fetal heart rate variability | Gestational week 28
  Fetal heart rate variability will be assessed by fMCG (fetal magnetocardiography).
Offsprings APGAR Score | Delivery
  APGAR of the newborn will be recorded at time of birth
Offsprings body weight | Delivery
  Body weight of the newborn will be recorded at time of birth
Offsprings body length | Delivery
  Length of the newborn will be recorded at time of birth
Offsprings head circumference | Delivery
  Head circumference of the newborn will be recorded at time of birth
Way of delivery | Delivery
  Way of delivery (cesarean section or vaginal delivery) will be documented
Time of delivery | Delivery
  Time of delivery will be recorded as gestational week

OTHER OUTCOMES:
Epigenetic modification | Delivery
  Effect of maternal glycaemia on epigenetic marks in cord blood leucocytes of the newborn will be investigated by analysing DNA methylation.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tuebingen, Department of Internal Medicine IV, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No
Due data protection regulation we will not be able to share patient level data.